CLINICAL TRIAL: NCT00825955
Title: A Randomized, Double-blind, Multi-center Phase III Study of Brivanib Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Subjects With Advanced Hepatocellular Carcinoma (HCC) Who Have Failed or Are Intolerant to Sorafenib: The BRISK PS Study (Brivanib Study in HCC Patients at Risk Post Sorafenib)
Brief Title: Comparison of Brivanib and Best Supportive Care to Placebo for Treatment of Liver Cancer for Those Subjects Who Have Failed Sorafenib Treatment
Acronym: BRISK PS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA182-034; EUDRACT #: 2008-005084-34
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — brivanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivanib (Experimental)
  Interventions: Drug: Brivanib; Procedure: Best Supportive Care
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo; Procedure: Best Supportive Care

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 800 mg, once daily, until disease progression or toxicity
  Other Names: BMS-582664
  Arms: Brivanib
Other: Placebo — Tablets, Oral, 0 mg, once daily, until disease progression or toxicity
  Arms: Placebo
Procedure: Best Supportive Care — Trans-Arterial Chemo-Embolization (TACE) Therapy

SUMMARY:
The purpose of this study is to determine if Brivanib is an effective treatment for liver cancer in patients who have failed or could not take Sorafenib

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Histologic or cytologic confirmed diagnosis of HCC
* Advanced disease defined as (i) disease not eligible for surgical or loco-regional therapy or (ii) disease progressive after surgical or loco-regional therapy
* Patient has failed ≥ 14 days of Sorafenib treatment
* Cirrhotic status of Child-Pugh Class A or B with a score of 7
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, 2
* Subjects who have a life expectancy of at least 8 weeks
* Adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* women of childbearing potential (WOCBP) who are unwilling or unable to use an acceptable method to avoid pregnancy
* Previous or concurrent cancer that is distinct in primary site
* History of active cardiac disease
* Thrombotic or embolic events within the past 6 months
* Any other hemorrhage/bleeding event > Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 within 4 weeks
* Inability to swallow tablets or untreated malabsorption syndrome
* History of human immunodeficiency virus (HIV) infection
* Prior use of systemic investigational agents for HCC (except for Sorafenib)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 587 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2011-11-15 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
To compare overall survival of subjects with advanced HCC who have progressed on/after or are intolerant to Sorafenib and receive Brivanib plus best supportive care (BSC) to those receiving placebo plus BSC | computerized tomography (CT)/ magnetic resonance imaging (MRI) every six weeks until progression or death

SECONDARY OUTCOMES:
To compare time to progression (TTP) (Investigator assessed using modified Response Evaluation Criteria In Solid Tumors (RECIST) for HCC criteria) | 35 months
To compare the Independent Radiological Review Committee (IRRC) assessed objective response rate (ORR) and disease control rate (DCR) using modified RECIST for HCC criteria | 35 months
To assess duration of response, duration of disease control and time to response | 6 weeks
To assess safety profile of brivanib. Safety will be assessed by the number of adverse events (AEs), serious adverse events (SAEs), periodic data monitoring committee (DMC) review | 35 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (102):
- United States (19):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Univ Of Ark For Med Sci, Little Rock, Arkansas
  - Loma Linda University Cancer Center, Loma Linda, California
  - Richard Finn, M.D., Los Angeles, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - UF Health Clinical Research Center, Gainesville, Florida
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - 3912 Taubman Center, Ann Arbor, Michigan
  - Henry Ford Health System Irb, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai School Of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Sci Univ, Portland, Oregon
  - University Of Pennsylvania, Philadelphia, Pennsylvania
  - University Of Texas, Houston, Texas
  - The University Of Texas Health Science Center, San Antonio, Texas
  - Mcguire Dvamc, Richmond, Virginia
- Argentina (2):
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
- Local Institution, Brussels, Belgium
- Brazil (4):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Salvador - Ba, Estado de Bahia
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo
- Canada (3):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario
- China (8):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Nanning, Guangxi
  - Local Institution, Wuhan, Hubei
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Tianjin, Tianjin Municipality
  - Local Institution, Hangzhou, Zhejiang
- France (11):
  - Local Institution, Bordeaux
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Lille
  - Local Institution, Lyon
  - Local Institution, Montpellier
  - Local Institution, Paris
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
  - Local Institution, Villejuif
- Germany (8):
  - Local Institution, Berlin
  - Local Institution, Frankfurt
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Halle
  - Local Institution, Hanover
  - Local Institution, Mainz
  - Local Institution, Ulm
  - Local Institution, Würzburg
- Greece (2):
  - Local Institution, Kifissia
  - Local Institution, Thessaloniki
- Local Institution, Hong Kong, Hong Kong
- India (4):
  - Local Institution, Kochi, Kerala
  - Local Institution, Chennai
  - Local Institution, Kolkata
  - Local Institution, New Delhi
- Italy (6):
  - Local Institution, Ancona
  - Local Institution, Meldola (fc)
  - Local Institution, Milan
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Pisa
- Japan (17):
  - Local Institution, Chiba, Chiba
  - Local Institution, Kashiwa-shi, Chiba
  - Local Institution, Ogaki-shi, Gifu
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Kochi, Kochi
  - Local Institution, Kyoto, Kyoto
  - Local Institution, Tsu, Mie-ken
  - Local Institution, Higashinari-ku, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Osaka-sayama-shi, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Bunkyo-ku, Tokyo
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Musashino-shi, Tokyo
  - Local Institution, Toyama, Toyama
  - Local Institution, Shimonoseki-shi, Yamaguchi
  - Local Institution, Nishinomiya-shi
- Mexico (3):
  - Local Institution, D.f., Mexico City
  - Local Institution, Cuernavaca, Morelos
  - Local Institution, Toluca, State of Mexico
- Local Institution, San Juan, Puerto Rico
- Local Institution, Moscow, Russia
- South Korea (4):
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
- Spain (3):
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Oviedo
- Taiwan (4):
  - Local Institution, Taichung
  - Local Institution, Tainan
  - Local Institution, Taipei
  - Local Institution, Taoyuan Hsien

REFERENCES:
- [Derived] Lencioni R, Montal R, Torres F, Park JW, Decaens T, Raoul JL, Kudo M, Chang C, Rios J, Boige V, Assenat E, Kang YK, Lim HY, Walters I, Llovet JM. Objective response by mRECIST as a predictor and potential surrogate end-point of overall survival in advanced HCC. J Hepatol. 2017 Jun;66(6):1166-1172. doi: 10.1016/j.jhep.2017.01.012. Epub 2017 Jan 26. PMID 28131794
- [Derived] Llovet JM, Decaens T, Raoul JL, Boucher E, Kudo M, Chang C, Kang YK, Assenat E, Lim HY, Boige V, Mathurin P, Fartoux L, Lin DY, Bruix J, Poon RT, Sherman M, Blanc JF, Finn RS, Tak WY, Chao Y, Ezzeddine R, Liu D, Walters I, Park JW. Brivanib in patients with advanced hepatocellular carcinoma who were intolerant to sorafenib or for whom sorafenib failed: results from the randomized phase III BRISK-PS study. J Clin Oncol. 2013 Oct 1;31(28):3509-16. doi: 10.1200/JCO.2012.47.3009. Epub 2013 Aug 26. PMID 23980090
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm